CLINICAL TRIAL: NCT00725049
Title: A Prospective, Multicenter, Randomized Multicenter Study of Short Implants Used to Obviate the Need for Sinus Augmentation: an Assessment of Clinical Outcomes and Resource Allocation.
Brief Title: An Evaluation of Integration Success and Maintenance of Short Implants in Maxillas Needing Sinus Augmentation
Acronym: Romeo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ZimVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2611
Record Dates: First submitted 2008-07-28; First posted 2008-07-30 (Estimated); Results first posted 2013-10-11 (Estimated); Last update posted 2024-02-20 (Actual); Status verified 2022-03

CONDITIONS: Tooth Disease; Partial Edentulism
Keywords: dental implants; Nanotite Certain implant; Osseotite; multicenter; randomized; clinical study; partial edentulism; crestal bone level; short fixed bridge; cost analysis
MeSH Terms: conditions — Tooth Diseases | interventions — Dental Implants

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dental implant (Nanotite) (Active Comparator): Dental implants of short length placed without sinus lifts
  Interventions: Device: Dental Implant (Nanotite)
- Control group (No Intervention): Dental implants of standard length placed simultaneously with sinus augmentation

INTERVENTIONS:
Device: Dental Implant (Nanotite) — Root form titanium dental implant
  Other Names: Nanotite
  Arms: Dental implant (Nanotite)

SUMMARY:
This prospective randomized study will evaluate the integration success while supporting a prosthesis for short implants placed into maxillary sites having minimal bone height that would otherwise need sinus augmentation. The resources utilized during treatment will be assessed.

Study (null) hypothesis: the overall benefit of using short length implants to avoid sinus augmentation procedures will offset differences in the cumulative implant survival rates observed between treatment groups.

DETAILED DESCRIPTION:
In this randomized study, patients needing restorations in the posterior maxilla will be randomly assigned to the short implant group (test) or the standard length and augmentation group (control). All implants will be placed using a two-stage approach with healing abutments placed at three months and temporary prosthesis at four months following implant and/ or sinus augmentation surgery. Time, materials, and efforts associated with treating test and control cases will be documented to allow an assessment of the costs incurred with each approach.

ELIGIBILITY:
Inclusion Criteria:

* patients of either sex and any race greater than 18 years of age
* patients with partial edentulism in the posterior maxilla requiring a unilateral implant-supported maxillary prosthesis
* patients with a residual alveolar floor of the sinus between 4 and 6 mm in height, as assessed on intraoral radiographs, and able to receive at least a 4mm wide implant
* patients must be physically able to tolerate conventional surgical and restorative procedures

Exclusion Criteria:

* patients with active infection or severe inflammation in the areas intended for implant placement
* patients with a > 10 cigarettes per day smoking habit
* patients with uncontrolled diabetes or metabolic bone disease
* patient with a history of therapeutic radiation to the head
* patients who are known to be pregnant
* patients with para-functional habits with evidence of severe bruxing or clenching
* patients not able to commit to a 3 year follow-up program

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2009-02 (Actual); Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mariano A Sanz, MD, DDS, Principal Investigator — Universidad Complutense de Madrid
Locations (1):
- Universidad Complutense de Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients enrolled in the study according to inclusion/ exclusion criteria as described in the protocol. Patient enrollment began February 2009 and ended February 2011. All study patients were enrolled at 3 European Universities (dental clinics).
Period: Overall Study
Arm/Group | Dental Implant (Nanotite) | Control Group
Started | 17 | 20
Completed | 17 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dental Implant (Nanotite) | Control Group | Total
Number analyzed (Participants) | 17 | 20 | 37
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 18 | 32
  >=65 years | 3 | 2 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 12 | 18
  Male | 11 | 8 | 19
Region of Enrollment [Number; unit: participants]
  Spain | 5 | 4 | 9
  Greece | 3 | 6 | 9
  Italy | 9 | 10 | 19

OUTCOME MEASURES:

1. Primary Outcome: Integration Success of Implant
Description: Number of enrolled and treated patients with integrated implants (no mobility detected) at time of analysis.
Time Frame: 3 years
Population: Number of participants used in analysis selected as per protocol
Measure: Number; unit: participants
Units Other Than Participants: Dental implants
Arm/Group | Dental Implant (Nanotite) | Control Group
Number analyzed (Participants) | 17 | 20
Number analyzed (Dental implants) | 31 | 35
participants | 17 | 20

ADVERSE EVENTS:
Time Frame: Adverse events are collected and reported from day 1 of the study to present time (entire duration of study).
Description: Adverse event data is collected by patient questioning and visual examination of patient's mouth during each study visit.
Arm/Group | Dental Implant (Nanotite) | Control Group
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/20
Other Adverse Events (participants affected / at risk) | 6/17 | 5/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dental Implant (Nanotite) (N=17) | Control Group (N=20)
Mobility (Surgical and medical procedures) | 6 (6) | 5 (5) — Dental implant mobility as detected by visual assessment,radiography, and patient complaint (symptoms).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI shall furnish SPONSOR with a copy of any proposed publication thirty (30) days prior to submission for publication for review and comment. SPONSOR may request PI to delay publishing such proposed publication for a maximum of an additional sixty (60) days in order to protect the potential patentability of any invention described therein.